CLINICAL TRIAL: NCT00451230
Title: Elucidating the Role of the Hypothalamic-Pituitary-Adrenal (HPA) Axis in the Mechanisms Underlying Cocaine Dependence
Brief Title: Metabolic Effects of Cocaine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: 2000p 000323; DA#14410
Record Dates: First submitted 2007-03-22; First posted 2007-03-23 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2002-10

CONDITIONS: Cocaine Dependence
Keywords: craving, insulin, leptin
MeSH Terms: conditions — Cocaine-Related Disorders; Insulin Resistance | interventions — Cocaine; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: cocaine
Drug: hydrocortisone

SUMMARY:
The goal of this this study is to elucidate the role of the HPA axis in the pathophysiology of cocaine dependence

ELIGIBILITY:
Inclusion Criteria:

* Individuals with DSM IV diagnosis of cocaine dependence, medically healthy

Exclusion Criteria:

* Other than cocaine dependence DSM-IV axis I diagnosis

Ages: 21 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15
Dates: Start 2005-06; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Igor Elman, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Rott D, Langleben DD, Elman I. Cocaine decreases plasma insulin concentrations in non-diabetic subjects: a randomized double-blind study. Diabet Med. 2008 Apr;25(4):510-1. doi: 10.1111/j.1464-5491.2008.02412.x. Epub 2008 Mar 13. No abstract available. PMID 18346162